CLINICAL TRIAL: NCT02254798
Title: Diagnostic and Prognostic Biomarkers for Acute Graft-versus-host Disease: a Prospective Single Centre Biological Study
Brief Title: Biomarkers for Acute Graft-versus-host Disease
Acronym: PLASMA-INCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI13015 PLASMA-INCA
Record Dates: First submitted 2014-09-17; First posted 2014-10-02 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Acute GVH Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample on day 7, 14, 21, 28 and at GVHD onset
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Transplanted patients: No intervention Prospective registration of patients receiving an allogeneic hematopoietic stem cell transplant
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — this is a non interventional study

SUMMARY:
Validation of already described biomarkers on acute GVHD prediction and severity Fecal calprotectin and alpha 1 anti-trypsin, plasmatic RER3a, IL-8, Elafin, TNFaR1, IL-2R alpha, HGF

DETAILED DESCRIPTION:
Description of the project: The main objective of this prospective biological single center study (non interventional) is to identify non invasive biomarkers able to diagnose acute GVHD and/or predict outcome of patients with acute GVHD. The primary objective of the study is double: (1): to evaluate markers as diagnostic markers of GVHD (2): to evaluate the potential of the markers as risk factor for steroid-refractory acute GVHD occurrence. Secondary objectives are: -to evaluate the markers as risk factors for GVHD -to evaluate the potential of these markers as prognostic factors of 6-month non-relapse mortality in patients with acute GVHD-to evaluate the additional value of the biomarkers to predict GVHD or steroid-refractory GVHD as compared to other known and routinely used risk factors (clinical grading system, performance status, albuminemia...). Stools and blood will be on day 7, 14, 21, 28 after transplantation and the first day of digestive GVHD. Management of patients will not differ from the usual care. Fecal calprotectin and alpha 1 anti-trypsin, plasmatic RER3a, IL-8, Elafin, TNFaR1, IL-2R alpha, HGF will be measured at each points by ELISA tests. 315 patients would be sufficient to estimate the area under the ROC curve with a half-width of the 99% confidence interval of 0.05, assuming 60% of patients would develop acute GVHD, and normally distributed markers. The diagnosis and prognosis values will be analyzed separately.

Expected results: If some biomarkers are found significantly associated with diagnosis or prognosis of acute GVHD, they will be compared with the current clinical, biological and histological markers. Indeed, these markers have a clinical potential impact only if they give similar or better information than routine currently available markers, ie: clinical GVHD grading system, performance status, gut endoscopy and histology. The non-invasivity of these biomarkers should also be taken into account (in comparison to histology).

Identification of diagnostic markers will avoid useless treatment with high dose corticosteroids in patients without GVHD Identification of prognostic markers will comfort the decision of a second-line treatment sooner than usually, ie: at GVHD onset. Indeed, the onset of a second-line treatment after a steroid-refractory GVHD varies from 3 to 21 days depending on clinical evolution of patients. If some prognostic markers are available at diagnosis, delay in second-line treatment can be shortened and the patient can consequently have an increased chance to response to an early treatment.

Identification of prognostic markers will also guide the corticosteroids decrease in patients with good prognosis GVHD

ELIGIBILITY:
Inclusion Criteria:

* adult patients receiving an allogeneic transplant
* informed consent signed

Exclusion Criteria:

* patient refusal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients receiving an allogeneic transplant
Sampling Method: Probability Sample
Enrollment: 315 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with an Acute Graft-versus-Host disease | The 6 first months after transplantation
  Evaluation of fecal and plasmatic markers as diagnostic markers of GVHD
Number of patients with an Acute Graft-versus-Host disease refractory to steroids | 14 days after acute graft-versus-host disease
  to evaluate the potential of these markers as risk factors for steroid-refractory acute GVHD occurrence

CONTACTS AND LOCATIONS:
Overall Officials: Marie Robin, Principal Investigator — Hôpital Saint-Louis
Locations (1):
- Hôpital Saint-Louis, Paris, France